CLINICAL TRIAL: NCT05648487
Title: A Phase II Study of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Combined With Sintilimab in Gastric Cancer With Peritoneal Metastasis
Brief Title: HIPEC Combined With Sintilimab for Gastric Cancer With Peritoneal Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-10
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Peritoneal Metastasis; HIPEC; PD1
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric Cancer With Peritoneal Metastasis, HIPEC, Anti-PD-1 Antibody (Experimental): 1. Surgical exploration, if PCI≤20, then we perform this study.
  2. HIPEC: HIPEC is performed after laparoscopic exploration, Mitomycin 30mg/m2, d1, Docetaxel 40mg/m2, d3, Oxaliplatin 65mg/m2, d5 within a week after surgical exploration;
  3. Chemotherapy(SOX) and anti-PD-1 antibody Sintilimab (Tyvyt®) treatment followed (4 cycles): SOX regimen: Oxaliplatin: 130 mg/m^2, IV, d1; S-1, 40-60 mg/m^2 bid, po, day 1-14, every 3 weeks for a total of 4 cycles; Sintilimab (Tyvyt®) 200mg fixed dose every 3 weeks, for a total of 4 cycles.
  4. Surgery: Imaging and secondary surgical exploration, assess the patient's condition and consider whether perform the cytoreductive surgery (resection of primary tumors and metastases ). After the surgery, HIPEC for three cycles, Mitomycin 30mg/m2, d1, Docetaxel 40mg/m2, d3, Oxaliplatin 65mg/m2, d5 within a week after surgery; For inoperable patients, continue to use standard chemotherapy.
  5. After the surgery, continue to use standard adjuvant chemotherapy.
  Interventions: Drug: HIPEC,anti-PD-1 antibody Sintilimab (Tyvyt®), Chemotherapy,Surgery

INTERVENTIONS:
Drug: HIPEC,anti-PD-1 antibody Sintilimab (Tyvyt®), Chemotherapy,Surgery — 1. HIPEC: HIPEC is performed after laparoscopic exploration, Mitomycin 30mg/m2, d1, Docetaxel 40mg/m2, d3, Oxaliplatin 65mg/m2, d5 within a week after surgical exploration.
  2. Chemotherapy(SOX) and anti-PD-1 antibody Sintilimab (Tyvyt®) treatment followed (4 cycles): SOX regimen: Oxaliplatin: 130 mg/m^2, IV, d1; S-1, 40-60 mg/m^2 bid, po, day 1-14, every 3 weeks for a total of 4 cycles; Sintilimab (Tyvyt®) 200mg fixed dose every 3 weeks, for a total of 4 cycles.
  3. Surgery: Imaging and secondary surgical exploration, assess the patient's condition and consider whether perform the cytoreductive surgery (resection of primary tumors and metastases). For patients undergoing surgery, HIPEC for three cycles followed, Mitomycin 30mg/m2, d1, Docetaxel 40mg/m2, d3, Oxaliplatin 65mg/m2, d5 within a week after surgery; For inoperable patients, continue to use standard chemotherapy of guidelines recommend.
  4. After the surgery, continue to use standard adjuvant chemotherapy.

SUMMARY:
To evaluate the Safety and Efficacy of HIPEC Combined With Sintilimab for Gastric Cancer Patients with Peritoneal Metastasis.

DETAILED DESCRIPTION:
Peritoneal metastasis is the most common pattern of disease relapse and is attributed to the dismal prognosis of the gastric cancer. The National Comprehensive Cancer Network (NCCN) guidelines suggest that systemic chemotherapy is the first-line standard strategy, and chemotherapy combined with trastuzumab for patients with positive HER-2. HIPEC can significantly improve survival in peritoneal metastasis from gastric cancer. PD-1/PD-L1 antibody has shown promising outcomes for unresectable or metastatic solid tumors. The present study aimed to evaluate the safety and efficacy of HIPEC combined with Sintilimab (Tyvyt®) in gastric cancer patients with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced gastric (gastroesophageal junction) adenocarcinoma confirmed by histology;
2. Age 18-75 years, Male or Non pregnant female
3. ECOG (Eastern Cooperative Oncology Group) : 0~1；
4. Negative for HER-2 by IHC/FISH；
5. Peritoneal metastasis is confirmed by laparoscopic exploration, and the PCI≤20；
6. Untreated (e.g. radiotherapy, chemotherapy, target therapy and immunotherapy);
7. Normal Bone marrow, liver and kidney function indices before the recruitment:
8. Expected survival≥ 12 week
9. Signed the Informed Consent Form, and blood and tissue samples can be obtained;

Exclusion Criteria:

1. Other distal metastases besides peritoneal metastases (e.g., liver, lung, pleural, brain, bone metastases, etc.);
2. Previous systemic therapy for gastric cancer;
3. Recurrent gastric cancer after surgery;
4. Cardiopulmonary dysfunction;
5. Immunosuppressive drugs(eg.Corticosteroids) were used within 14 days before treatment, eg.corticosteroids,
6. There is any active autoimmune disease or a history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma in childhood have been completely relieved, and those who do not need any intervention after adulthood can be included Asthma requiring medical intervention with bronchodilator was not included.)
7. Allergy to the drugs in this protocol；
8. Patients with other diseases not suitable for inclusion, such as immune deficiency, active tuberculosis, hepatitis B (non-active hepatitis B surface antigen (HBsAg) carriers, hepatitis B virus titer <500IU/ml after treatment and with normal liver function can be included), hepatitis C virus positive;
9. A history of idiopathic pulmonary fibrosis, tissue pneumonia, drug pneumonia, idiopathic pneumonia, or r active pneumonia;
10. Other patients who were considered unsuitable for inclusion by the researchers;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection | 3 months
  the rate of R0 resection

SECONDARY OUTCOMES:
Overall survival time | 2 years
  Overall survival time(OS) refers to the time of first use of the drug to the time of death. At the end of the study, if the subject is still alive, refer the known "date of last survival of the subject" as the date of censoring.
ORR | 3 months
  Objective response rate(ORR): ORR = (number of subjects with complete response (CR) + partial response (PR))/total number of subjects ×100%. Measurable lesion according to the RECISTv1.1
Event-Free Survival | 2 years
  Defined as the interval between the first conversion therapy and the first recorded related events, including preoperative disease progression, postoperative disease recurrence, and death from any cause.
Relapse-Free Survival | 2 years
  Defined as postoperative the first recorded postoperative recurrence of disease or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Cui, Doctor, Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Batran SE, Homann N, Pauligk C, Illerhaus G, Martens UM, Stoehlmacher J, Schmalenberg H, Luley KB, Prasnikar N, Egger M, Probst S, Messmann H, Moehler M, Fischbach W, Hartmann JT, Mayer F, Hoffkes HG, Koenigsmann M, Arnold D, Kraus TW, Grimm K, Berkhoff S, Post S, Jager E, Bechstein W, Ronellenfitsch U, Monig S, Hofheinz RD. Effect of Neoadjuvant Chemotherapy Followed by Surgical Resection on Survival in Patients With Limited Metastatic Gastric or Gastroesophageal Junction Cancer: The AIO-FLOT3 Trial. JAMA Oncol. 2017 Sep 1;3(9):1237-1244. doi: 10.1001/jamaoncol.2017.0515. PMID 28448662
- [Background] Okabe H, Ueda S, Obama K, Hosogi H, Sakai Y. Induction chemotherapy with S-1 plus cisplatin followed by surgery for treatment of gastric cancer with peritoneal dissemination. Ann Surg Oncol. 2009 Dec;16(12):3227-36. doi: 10.1245/s10434-009-0706-z. Epub 2009 Sep 24. PMID 19777180
- [Background] Ishigami H, Fujiwara Y, Fukushima R, Nashimoto A, Yabusaki H, Imano M, Imamoto H, Kodera Y, Uenosono Y, Amagai K, Kadowaki S, Miwa H, Yamaguchi H, Yamaguchi T, Miyaji T, Kitayama J. Phase III Trial Comparing Intraperitoneal and Intravenous Paclitaxel Plus S-1 Versus Cisplatin Plus S-1 in Patients With Gastric Cancer With Peritoneal Metastasis: PHOENIX-GC Trial. J Clin Oncol. 2018 Jul 1;36(19):1922-1929. doi: 10.1200/JCO.2018.77.8613. Epub 2018 May 10. PMID 29746229
- [Background] Yang XJ, Huang CQ, Suo T, Mei LJ, Yang GL, Cheng FL, Zhou YF, Xiong B, Yonemura Y, Li Y. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy improves survival of patients with peritoneal carcinomatosis from gastric cancer: final results of a phase III randomized clinical trial. Ann Surg Oncol. 2011 Jun;18(6):1575-81. doi: 10.1245/s10434-011-1631-5. Epub 2011 Mar 23. PMID 21431408
- [Background] Jiang H, Yu X, Li N, Kong M, Ma Z, Zhou D, Wang W, Wang H, Wang H, He K, Li Z, Lu Y, Zhang J, Zhao K, Zhang Y, Xu N, Li Z, Liu Y, Wang Y, Wang Y, Teng L. Efficacy and safety of neoadjuvant sintilimab, oxaliplatin and capecitabine in patients with locally advanced, resectable gastric or gastroesophageal junction adenocarcinoma: early results of a phase 2 study. J Immunother Cancer. 2022 Mar;10(3):e003635. doi: 10.1136/jitc-2021-003635. PMID 35296556
- [Background] Bonnot PE, Piessen G, Kepenekian V, Decullier E, Pocard M, Meunier B, Bereder JM, Abboud K, Marchal F, Quenet F, Goere D, Msika S, Arvieux C, Pirro N, Wernert R, Rat P, Gagniere J, Lefevre JH, Courvoisier T, Kianmanesh R, Vaudoyer D, Rivoire M, Meeus P, Passot G, Glehen O; FREGAT and BIG-RENAPE Networks. Cytoreductive Surgery With or Without Hyperthermic Intraperitoneal Chemotherapy for Gastric Cancer With Peritoneal Metastases (CYTO-CHIP study): A Propensity Score Analysis. J Clin Oncol. 2019 Aug 10;37(23):2028-2040. doi: 10.1200/JCO.18.01688. Epub 2019 May 14. PMID 31084544